CLINICAL TRIAL: NCT06992284
Title: A Prognostic Study Using Health Insurance Claim for Patients With Cardiovascular Disease in Niigata
Brief Title: A Prognostic Study for Patients With Cardiovascular Disease in Niigata
Status: Enrolling by invitation | Type: Observational
Sponsor: Niigata University Medical & Dental Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0250
Record Dates: First submitted 2025-03-05; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to investigate the prognosis of cardiovascular disease in Niigata Prefecture.

Specifically, it aims to clarify the current status of medical treatment for cardiovascular disease patients in regional cities in Japan, where the population is aging.

With patient consent, the study will track long-term medical treatment progress using health insurance claim data recorded in Japan's unique social security system.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 or older at the time of enrollment (regardless of gender).
* Individuals who have been hospitalized in the cardiology department of a participating medical institution.
* Individuals covered by Japan's National Health Insurance (NHI) or the Late-stage Elderly Medical Care System, which provide health coverage for self-employed individuals, retirees, and the elderly.

Exclusion Criteria:

* Individuals who are unable to obtain consent from themselves or their legally authorized representatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants are individuals aged 18 or older who have been hospitalized in the cardiology department of a participating medical institution and are covered by Japan's National Health Insurance or the Late-stage Elderly Medical Care System
Sampling Method: Probability Sample
Enrollment: 8500 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2047-12-31 (Estimated); Study Completion 2050-05 (Estimated)

PRIMARY OUTCOMES:
The rate of deterioration in care dependency levels as defined by Japan's Long-Term Care Insurance system | through study completion, an average of 1 year
  through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Niigata University, Niigata, Niigata, Japan